CLINICAL TRIAL: NCT06632574
Title: A Phase I Clinical Study Evaluating the Safety, Tolerability, and Pharmacokinetic Characteristics of Paclitaxel Cationic Liposome for Injection in the Treatment of Patients With Advanced Solid Tumors Via Transcatheter Arterial Infusion Therapy.
Brief Title: A Clinical Study of Paclitaxel Cationic Liposomes for the Treatment of Patients With Advanced Solid Tumors
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: CSPC ZhongQi Pharmaceutical Technology Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HA131-003
Record Dates: First submitted 2024-09-27; First posted 2024-10-09 (Actual); Last update posted 2024-10-09 (Actual); Status verified 2024-10

CONDITIONS: Advanced Solid Tumor

STUDY DESIGN:
Intervention Model Description: All participants receive the same treatment, and there is no comparison group.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Experimental arm (Experimental): Patients with advanced solid tumors received arterial infusion chemotherapy with paclitaxel cationic liposomes, at a dosage range of 33 mg/m^2 to 66 mg/m^2.
  Interventions: Drug: paclitaxel cationic liposomes

INTERVENTIONS:
Drug: paclitaxel cationic liposomes — Paclitaxel cationic liposomes is a modified new drug. In this study, administration is performed through arterial catheter infusion.

SUMMARY:
This is an open-label, dose-escalation and expansion, cohort expansion, multicenter Phase I clinical study in patients with advanced solid tumors.

DETAILED DESCRIPTION:
This is an open-label, dose-escalation and expansion, cohort expansion, multicenter Phase I clinical study in patients with advanced solid tumors.

The study aims to evaluate the safety, tolerability, pharmacokinetic characteristics, and preliminary efficacy of paclitaxel cationic liposomes for injection administered via transcatheter arterial infusion in the treatment of advanced solid tumors.

Paclitaxel cationic liposomes will be administered via arterial infusion on the first day of each cycle, with each treatment cycle lasting 3 weeks. Eligible participants will receive 4-6 cycles of study treatment. Treatment may be terminated early in the event of the following: disease progression, intolerable toxicity, initiation of new anti-tumor therapy, withdrawal of informed consent, loss to follow-up, death, or any other circumstances meeting the criteria for treatment discontinuation (whichever occurs first).

ELIGIBILITY:
Inclusion Criteria:

* 1. Age ≥ 18 years.
* 2. Histologically or cytologically diagnosed advanced solid tumors suitable for arterial infusion chemotherapy, including but not limited to the following types:

  * Gastrointestinal tumors (e.g., gastric cancer, liver cancer, cholangiocarcinoma, pancreatic cancer, colorectal cancer, etc.);
  * Gynecological tumors (e.g., ovarian cancer, endometrial cancer, etc.);
  * Non-small cell lung cancer (NSCLC);
  * Liver metastases.
* 3. According to RECIST 1.1, at least one measurable lesion in the arterial infusion area.
* 4. If life-threatening primary lesions are within the arterial infusion area, limited lesions outside the arterial infusion area at baseline are acceptable.
* 5. Eastern Cooperative Oncology Group (ECOG) performance status score of 0-2.
* 6. Life expectancy of at least 3 months.
* 7. Adequate organ function, with laboratory tests meeting the following criteria (no blood transfusion or hematopoietic growth factors within 14 days):

  * Absolute neutrophil count (ANC) ≥ 1.5 × 10^2/L.
  * Platelets (PLT) ≥ 100 × 10^9/L.
  * Hemoglobin (Hb) ≥ 90 g/L.
  * Total bilirubin (TBIL) ≤ 1.5 × upper limit of normal (ULN); for individuals with liver metastasis or liver cancer, TBIL ≤ 2 × ULN.
  * Alanine aminotransferase (ALT), aspartate aminotransferase (AST) ≤ 2.5 × ULN; for liver metastasis or liver cancer, ALT, AST ≤ 5 × ULN.
  * Creatinine clearance (Ccr) > 50 mL/min (calculated using the Cockcroft-Gault formula).
  * Activated partial thromboplastin time (APTT) ≤ 1.5 × ULN; international normalized ratio (INR) ≤ 1.5 × ULN.
* 8. Fertile individuals (male and female) must agree to use reliable contraceptive methods (hormonal contraceptives, barrier methods, or abstinence) with their partners during the trial and for at least 6 months after the last dose of study medication. Women of childbearing potential must have a negative pregnancy test within 7 days prior to enrollment.
* 9. Fully understand the clinical trial and voluntarily sign a written informed consent form.

Exclusion Criteria:

* 1. Received chemotherapy, radiotherapy, biological therapy, endocrine therapy, targeted therapy, immunotherapy, or participated in another clinical trial within 4 weeks prior to the first administration of the study drug, or within 4 weeks or 5 half-lives of the treatment drug (whichever is shorter).
* 2. Known symptomatic central nervous system or meningeal metastases, or other evidence of uncontrolled central nervous system or meningeal metastases, deemed unsuitable for enrollment by the investigator.
* 3. Unresolved adverse reactions from previous anti-tumor treatments not yet recovered to CTCAE 5.0 grade ≤ 1 (except for alopecia or other toxicities deemed non-risky by the investigator).
* 4. Concurrent participation in another clinical trial, unless it is observational (non-interventional) or in the follow-up period of an interventional trial.
* 5. Major surgery or invasive intervention within 28 days prior to the first dose.
* 6. Use of any anti-cancer herbal or traditional Chinese medicine approved by the National Medical Products Administration (NMPA) within 14 days prior to the first dose.
* 7. Known severe allergic reactions to the study drug or its components/excipients.
* 8. Active bacterial, fungal, or viral infections requiring intravenous antibiotic, antifungal, or antiviral treatment prior to the first dose. Participants receiving prophylactic infection treatment with no signs of active infection may be considered for enrollment.
* 9. History of immunodeficiency diseases, including positive HIV antibodies.
* 10. Hepatitis B surface antigen (HBsAg) positive with HBV DNA above the measurable limit or 1000 copies/mL (500 IU/mL) (whichever is lower), or HCV antibody positive with HCV RNA above the measurable limit or 1000 copies/mL (whichever is lower). Individuals whose levels are reduced to below the standard following antiviral treatment may be screened.
* 11. Underlying medical conditions (including laboratory abnormalities), alcohol or drug abuse, or dependence that may impair the administration of study drugs or interpretation of drug toxicity and adverse events (AEs), or lead to insufficient or reduced trial compliance.
* 12. Severe cardiovascular disease history, including but not limited to:

  * Severe cardiac rhythm or conduction abnormalities requiring clinical intervention, such as ventricular arrhythmias or grade II-III atrioventricular block;
  * Average QTcF > 450 ms from three resting 12-lead ECGs;
  * Acute coronary syndrome, congestive heart failure, stroke, or other grade 3 or higher cardiovascular events within 6 months prior to the first dose;
  * New York Heart Association (NYHA) class II or higher, or left ventricular ejection fraction (LVEF) < 50%;
  * Any factors increasing the risk of QTc prolongation or arrhythmias, such as heart failure, hypokalemia, congenital long QT syndrome, family history of long QT syndrome or unexplained sudden death in a first-degree relative under 40 years old, or concurrent use of QT-prolonging drugs.
  * Uncontrolled hypertension (screening systolic BP ≥ 160 mmHg and/or diastolic BP ≥ 100 mmHg).
* 13.History of other malignancies within the past 3 years or concurrent active malignancies (localized, curable malignancies such as basal cell carcinoma of the skin, squamous cell carcinoma of the skin, superficial bladder cancer, in situ prostate cancer, cervical carcinoma in situ, and in situ breast cancer may be included).
* 14. Patients with ultrasound-detected limb vascular thrombosis with potentially serious consequences during screening, or participants with thromboembolic events within 3 months prior to enrollment.
* 15. Individuals with coagulopathy or a history of severe bleeding, or who experienced major bleeding events such as intracranial hemorrhage, gastrointestinal bleeding, or purpura within the last 3 months.
* 16. Pregnant or breastfeeding women.
* 17. Any other reasons deemed by the investigator to make the individual unsuitable for participation in the clinical trial.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2014-03-19 (Actual); Primary Completion 2025-10-31 (Estimated); Study Completion 2027-03-31 (Estimated)

PRIMARY OUTCOMES:
The incidence of dose-limiting toxicity (DLT) | At the end of Cycle 1 ( each cycle is 21 days)
Incidence and severity of Adverse Events (AEs) and Serious Adverse Events (SAEs)(according to NCI-CTCAE 5.0) | Up to approximately 3 years

SECONDARY OUTCOMES:
AUC0-t | At the end of Cycle 4 ( each cycle is 21 days)
AUC0-∞ | At the end of Cycle 4 ( each cycle is 21 days)
Cmax | At the end of Cycle 4 ( each cycle is 21 days)
Kel | At the end of Cycle 4 ( each cycle is 21 days)
Tmax | At the end of Cycle 4 ( each cycle is 21 days)
Vd | At the end of Cycle 4 ( each cycle is 21 days)
t1/2 | At the end of Cycle 4 ( each cycle is 21 days)
CL | At the end of Cycle 4 ( each cycle is 21 days)
Overall response rate (ORR) | Up to approximately 3 years
Disease control rate (DCR) | Up to approximately 3 years
Duration of Response (DoR) | Up to approximately 3 years
Progression-Free-Survival (PFS) | Up to approximately 3 years
Overall survival (OS) | Up to approximately 3 years

CONTACTS AND LOCATIONS:
Locations (1):
- Zhongda Hospital, Southeast University, Nanjing, China